CLINICAL TRIAL: NCT02845973
Title: Study of Fecal Bacteria in Early Diagnosis of Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai 10th People's Hospital (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Jing-yuan Fang, MD, Ph. D, Chief, Division of Gastroenterology and Hepatology, Shanghai Jiao Tong University School of Medicine
Other Study IDs: RJ20160701
Record Dates: First submitted 2016-07-17; First posted 2016-07-27 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Colorectal Neoplasms
Keywords: gut microbiota
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Gastrointestinal Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — feces of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- test cohort: The test cohort was from Fudan University Shanghai Cancer Center (August 2016 to December 2016) and ECRJ-East Campus of Renji hospital (January 2012 to March 2017);
  Interventions: Biological: gut microbiota
- validation cohort: The validation cohort was from Shanghai Tenth People's Hospital (October 2015 to November 2016) and WCRJ-West Campus of Renji hospital (July 2016 to March 2017)
  Interventions: Biological: gut microbiota

INTERVENTIONS:
Biological: gut microbiota

SUMMARY:
The aim of the study is to identify and verify one or more gut bacteria of which the abundance in feces may help to early diagnosis colorectal cancer.

DETAILED DESCRIPTION:
Gut microbiota is closely related to human gut neoplasm. According to recent statistics, the abundance of FN (Fusobacterium Nucleatum) is connected with the development and progression of CRCs (colorectal cancers). Subsequent research shows identifying multiple microbial-specific genes in human feces using qPCR (quantitative Polymerase Chain Reaction) may help diagnosis of early stage colorectal cancer. Currently little is known about the relationship between single abundance of specific gut microbiota and colorectal cancer in different stage. Moreover, finding early-stage CRCs is still of great challenge partially due to precancerous diseases like colorectal adenoma which remain difficult to differentiate from early-stage CRC under endoscope. Conventional clinic methods predicting CRCs largely depend on serum CEA (serum Carcino Embryonic Antigen) and OB(fecal occult blood test), which lack of adequate sensitivity and specificity especially in early stage CRCs. The investigators' work focuses on the abundance of gut microbiota in feces from people with colon neoplasm and its comparison with classical indicators such as CEA and OB, aiming to reveal and testify its potential role on assisting diagnosis of CRCs in different stage as a none-invasive cost-effective method.

ELIGIBILITY:
Inclusion Criteria:

* Patients age from 40 to 85 years old
* Patients with endoscopic or pathological confirmed healthy, adenoma, inflammation, early or late stage of colorectal cancer
* Patients with valid CEA(carcino embryonic antigen) and OB(occult blood) test result in 1 year before or after the coloscopy or surgery

Exclusion Criteria:

* Patients with history of colorectal cancer
* Patients with long term use of antibiotics or probiotics
* Patients with uncontrolled diabetes, hypertension or hepatitis
* Patients with a history of subtotal gastrectomy or partial bowel resection
* Patients who are not able to cooperate
* Patients with medical conditions who are not appropriate to participate the study
* Patients who are taking aspirin, NSAIDs (nonsteroidal antiinflammatory drugs), COX2(cyclo-oxygen-ase 2) inhibitors.

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese people
Sampling Method: Non-Probability Sample
Enrollment: 1325 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
differences in abundance of gut microbiota | 1 year
  differences in abundance of gut microbiota for participants with different clinical outcomes confirmed by qPCR(quantitive polymerase chain reaction)

SECONDARY OUTCOMES:
evidence of colorectal neoplasia | 1 year
  Different outcomes for colorectal neoplasia confirmed by coloscopy

OTHER OUTCOMES:
diet difference in patients with different clinical outcomes | 1 year
  Diet difference in patients with different clinical outcomes by a food-frequency questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Institute of Digestive Disease, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xie YH, Gao QY, Cai GX, Sun XM, Sun XM, Zou TH, Chen HM, Yu SY, Qiu YW, Gu WQ, Chen XY, Cui Y, Sun D, Liu ZJ, Cai SJ, Xu J, Chen YX, Fang JY. Fecal Clostridium symbiosum for Noninvasive Detection of Early and Advanced Colorectal Cancer: Test and Validation Studies. EBioMedicine. 2017 Nov;25:32-40. doi: 10.1016/j.ebiom.2017.10.005. Epub 2017 Oct 4. PMID 29033369